CLINICAL TRIAL: NCT07136051
Title: Evaluation of the Survival of Fissure Sealants Applied With Different Pretreatment Methods on Permanent First Molars: A One-Year Follow-Up
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Handan Vural (Other)
Collaborators: Inonu University (Other)
Responsible Party: Sponsor-Investigator, Handan Vural, Assistant Professor, Inonu University
Organization: Inonu University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 7706
Record Dates: First submitted 2025-08-19; First posted 2025-08-22 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Fissure Sealant; Deproteinization; Bonding Agent; Molar Teeth; Etching
Keywords: fissure sealant; deproteinization; bonding agent; etching

STUDY DESIGN:
Intervention Model Description: In this split-mouth design study, at least three fully erupted permanent molars from each participant will be included. The teeth will be randomly allocated into groups, and fissure sealants will be applied with the appropriate pretreatments according to the assigned group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A: Acid etching + sealant (Active Comparator): Sealant application is a preventive conservative approach involving the introduction of sealants into the pits and fissures of caries prone teeth; this sealant then bonds to the tooth micromechanically, providing a physical barrier that keeps bacteria away from their source of nutrients. Acid pretreatment of the enamel to enhance retention is considered a standard procedure prior to the application of resin-based fissure sealants. Currently, the most commonly used phosphoric acid concentrations are 35% and 37%.
  Interventions: Procedure: Ethcing; Procedure: Application of resin-based fissure sealant
- Group B: Acid etching + deproteinization + sealant (Active Comparator): The use of phosphoric acid is a well-accepted, conventional method used to create micro-porosities, which are the key in providing sealant retention. However, organic remnants as well as fissure morphology and aprismatic enamel structure can decrease etching ability and thus prevent adequate adhesion.Conventional phosphoric acid can only demineralize the inorganic component of enamel and cannot completely remove the protein content within the enamel. Some proteins are also embedded within the enamel crystals. The inadequate penetration of resin into enamel may also result from the Type 3 etching pattern observed after conventional etching. Studies have shown that after using sodium hypochlorite to remove enamel proteins, Type 1 and Type 2 etching patterns are more frequently observed. The literature indicates that the enamel deproteinization technique with sodium hypochlorite is an effective method for removing organic material from the occlusal enamel surfaces of teeth.
  Interventions: Procedure: Ethcing; Procedure: Deproteinization; Procedure: Application of resin-based fissure sealant
- Group C: Acid etching + bonding agent + sealant (Active Comparator): Various methods for preparing fissures, such as pumice prophylaxis, bonding agents, lasers, air abrasion, and sodium hypochlorite deproteinization, have been recommended to improve sealant retention The use of adhesive systems prior to fissure sealant application had a positive effect on increasing penetration and improving the retention rate. It also appears that the use of bonding-agents that involve a separate acid-etching step (fourth and fifth generations) provides better sealant retention than self-etching adhesives (sixth and seventh generations).
  Interventions: Procedure: Ethcing; Procedure: Bonding; Procedure: Application of resin-based fissure sealant

INTERVENTIONS:
Procedure: Ethcing — Etching: After polishing all teeth included in the study with a polishing brush, Vococid (Voca, Germany) etching gel will be applied to the surface and left for 15 seconds, then rinsed and dried.
Procedure: Deproteinization — The teeth randomly assigned to Group B will receive 5.25% NaOCl applied with a sterile cotton pellet for 60 seconds after acid etching, followed by rinsing and drying.
  Arms: Group B: Acid etching + deproteinization + sealant
Procedure: Bonding — The teeth randomly assigned to Group C will receive Futurabond® M+ (Voco, Germany) applied with a brush following acid etching. After gently drying with air for 5 seconds, the bonding step will be completed by light-curing for 10 seconds.
  Arms: Group C: Acid etching + bonding agent + sealant
Procedure: Application of resin-based fissure sealant — After completing the pretreatment steps for all groups, Grandio Seal (Voco GmbH, Germany) will be applied to the pits and fissures on the tooth surface and light-cured for 20 seconds. The procedure will be completed after checking the surface.

SUMMARY:
Objective:

This study aims to evaluate the effect of two different pretreatment protocols-enamel deproteinization and bonding agent application-on the one-year survival of fissure sealants applied to permanent first molars in children.

Background:

Dental caries is a preventable yet highly prevalent multifactorial disease. Deep pits and fissures are particularly susceptible to caries development, especially in newly erupted molars. Although fissure sealants are considered one of the most effective preventive methods, their clinical success is largely dependent on long-term retention. Contamination of etched enamel surfaces with saliva or gingival fluid is a primary cause of sealant failure. To improve sealant adhesion, several pretreatment methods have been suggested, including bonding agents and enamel deproteinization.

Methods:

This randomized, controlled, double-blind clinical trial with a split-mouth design was conducted on healthy children aged 7-14 years. Each child contributed at least three permanent first molars to the study, randomly assigned to one of three groups:

Group A - Acid etching + sealant; Group B - Acid etching + deproteinization + sealant; Group C - Acid etching + bonding agent + sealant. Clinical evaluations were performed at 3, 6, and 12 months using visual and tactile methods. Sealant retention, caries incidence, and marginal discoloration were recorded based on standardized criteria.

Results & Conclusion:

This study seeks to clarify whether bonding agent or deproteinization pretreatment significantly improves sealant retention and reduces caries incidence compared to the conventional approach. Findings may contribute to defining the most effective clinical protocol for fissure sealant application, ultimately enhancing caries prevention and long-term treatment success in pediatric dental care.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children aged 8-15 years.
* Fully erupted or completely impacted teeth that are clinically and radiographically confirmed to be caries-free or present with demineralized fissures scored as ICDAS 1-2.
* Children demonstrating cooperative behavior, with a Frankl Behavior Rating Scale score of 3 or 4.
* Oral Hygiene Index (OHI-S) score ≤ 3
* Written informed consent obtained from the parent or legal guardian.

Exclusion Criteria:

* Partially erupted second permanent molars
* Teeth presenting with severe hypoplasia, hypomineralization, extensive restorations, or cavitated carious lesions.
* History of systemic disease or long-term medication use.
* Known allergy to resin-based or glass ionomer materials.
* Presence of parafunctional habits.

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-08-03 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Modified Simonsen Criteria | Follow-up appointments were scheduled for children at 3, 6, and 12 months following the initial treatment.
  Score 0 Fissure sealant is completely in the mouth and there is no new caries. Score 1 Partial loss of fissure sealant, no new caries. Score 2 Partial loss of fissure sealant and new caries. Score 3 Complete loss of fissure sealant, no new caries. Score 4 Complete loss of fissure sealant and new caries
Edge Integrity Evaluation Criteria | Follow-up appointments were scheduled for children at 3, 6, and 12 months following the initial treatment
  0: The fissure sealant and tooth surface are intact and cannot be distinguished with a probe. 1: The edges of the fissure sealants can be distinguished with a probe. 2: There is a gap along the edge of the fissure sealant and deep cracks reaching the central fossa
Marginal Coloration Evaluation Criteria | Follow-up appointments were scheduled for children at 3, 6, and 12 months following the initial treatment.
  0 No color change between fissure sealant and tooth. 1:Color change in only one area. 2:Color change in many areas. 3:Severe color change indicating leakage.
Anatomical Form Evaluation Criteria | Follow-up appointments were scheduled for children at 3, 6, and 12 months following the initial treatment.
  0 Consistent with and continuous with occlusal form and structure. 1 Change in anatomical form but all pits and fissures covered. 2a Partial loss of one or two pits or fissures but no need to repair or replace fissure sealant. 2b Partial loss of pits and fissures, fissure sealant needs to be replaced or repaired. 3 Loss of all pits and fissures. 7 Partial loss due to occlusion 9 Bleb not connected to margins

CONTACTS AND LOCATIONS:
Overall Officials: handan vural, Assistant Professor, Study Chair — Department of Pediatric Dentistry, Faculty of Dentistry, Inonu University
Locations (1):
- Department of Pediatric Dentistry, Faculty of Dentistry, Inonu University, Battalgazi, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
IPD used in the results publication
Supporting Information: Study Protocol, CSR
Time Frame: Beginning 6 months and ending 1 years after the publication of results
Access Criteria: Access to individual participant data (IPD) and supporting materials will be made available to qualified researchers upon reasonable request. The following details apply:
  Who can access the data: Qualified academic researchers with a valid scientific purpose.
  What can be accessed: De-identified IPD, study protocol, statistical analysis plan, informed consent forms, and ethics approval documents.
  How to access: Interested researchers must submit a written request, including a brief research proposal and documentation of ethics committee approval. Requests should be sent to the corresponding author via email. Data sharing will be conducted in accordance with ethical guidelines and applicable data protection regulations.

REFERENCES:
- [Background] Khare M, Suprabha BS, Shenoy R, Rao A. Evaluation of pit-and-fissure sealants placed with four different bonding protocols: a randomized clinical trial. Int J Paediatr Dent. 2017 Nov;27(6):444-453. doi: 10.1111/ipd.12281. Epub 2016 Dec 26. PMID 28024165
- [Background] Nair SM, Nene KS, Tirupathi S, Mathur AA, Khan HA, Godbole NM, Patil PP, Deolikar SA. Effect of Enamel Deproteinization Prior to Etching on the Clinical Performance of Resin-based Pit and Fissure Sealants: A Split-mouth Double-blinded Pilot Randomized Controlled Trial. Int J Clin Pediatr Dent. 2025 Feb;18(2):119-125. doi: 10.5005/jp-journals-10005-3051. Epub 2025 Mar 20. PMID 40417445